CLINICAL TRIAL: NCT01697891
Title: Effectiveness of Acupuncture-like Transcutaneous Nerve Stimulation (ALTENS) in Improving Dysphagia and Associated Symptoms of Chemotherapy and/or Intensity Modulated Radiation Therapy (IMRT) for Head and Neck Cancers: A Pilot Study
Brief Title: A Pilot Study of ALTENS in Improving Dysphagia Induced by IMRT for Head and Neck Cancers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Raimond Wong, Associate Professor, Department of Oncology, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MU12-530
Record Dates: First submitted 2012-09-26; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Head and Neck Cancer; Dysphagia
Keywords: Radiation Treatment; Head and Neck Cancer; Dysphagia
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALTENS (Experimental): Patients in this arm will be treated with Acupuncture-like Transcutaneous Electrical Nerve Stimulation using Codetron (Codetron ALTENS)
  Interventions: Device: Codetron ALTENS

INTERVENTIONS:
Device: Codetron ALTENS — ALTENS stimulation of a set of selected acupuncture points for 20 minutes in each treatment. Two treatments per week for a total of 12 treatments to be delivered within 8 weeks.

SUMMARY:
Study hypothesis: ALTENS techniques, administered within the first 3 months after radiation completion, can improve radiation-induced dysphagia and associated symptoms in head and neck cancer patients. This beneficial effect is mediated by the reduction of chronic inflammatory response of swallowing musculature to radiation, consequently a reduction in muscle fibrosis.

Primary study objective: To evaluate the effectiveness of ALTENS in relieving radiation-induced dysphagia. Eating Assessment Tool (EAT-10) scores will be used for this primary study endpoint.

DETAILED DESCRIPTION:
Difficulty in swallowing is a concerning symptom after radiation treatment for some types of head and neck cancers. Swallowing becomes difficult when radiation damage induces inflammation (with swelling and pain) in the inner covering tissues of the throat and muscles that involve in the swallowing process. Currently, supportive measures are used to manage this symptom while waiting for the tissue damages to heal. In some patients, the inflamed muscles develop scar tissues causing long-term swallowing difficulty and narrowing of the swallowing passage. Needle acupuncture may help to reduce tissue inflammation and may lessen the severity of swallowing difficulty. However, needle puncture is often not desired by patients. Acupuncture-like transcutaneous electrical nerve stimulation (ALTENS) is like acupuncture treatment, but the acupuncture points are stimulated with mild electrical stimulation without needles, simplifying treatment delivery. This study is to examine if a pre-selected set of acupuncture points treated using ALTENS can reduce swallowing difficulty. There will be a total of 12 treatments given over 6 to 8 weeks. Changes in severity of swallowing difficult after treatment will be assessed using 2 subjective assessment tools.

ELIGIBILITY:
Inclusion Criteria:This study will recruit patients with head and neck cancers treated with radiation+/- chemotherapy and who meet the following criteria (EAT-10 assessment will be used for screening):

Inclusion Criteria

1. present with dysphagia symptoms
2. with no evidence of residue cancer
3. are within 3 months (but past 1 month) after treatment completion
4. show positive dysphagia (EAT-10 score of > 3) and/ or aspiration on barium swallow study
5. are over 18 years old
6. are able to read and write fluent English
7. can give informed consent

Exclusion Criteria:

1. have unstable heart disease
2. have infectious disease transmissible by blood or body fluid, including hepatitis and HIV
3. have skin disease at site of study acupuncture points that prevents the application of electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in Subjective Dysphagia Assessment Score: EAT-10 from baseline | 3 months after treatment completion
  EAT-10 is a self-administered questionnaire for subjective assessment of dysphagia. It consists of 10 items and each item is scored using a 5-point Likert scale. The higher the point, the more severe the problem being scored. Normative data suggested that a total score of 3 or higher is abnormal.

SECONDARY OUTCOMES:
Change in M. D. Anderson dysphagia inventory from baseline | 3 months after treatment completion
  M. D. Anderson dysphagia inventory (MDADI) is a self-administered questionnaire designed specifically to assess the quality of life for head and neck cancer patients who suffer from dysphagia. It incorporated three domains: emotional, functional and physical, and one global question. There are a total of 20 items.Each item is scored on a scale of 1 to 5 with 1 being strongly agree and 5 strongly disagree except for two items, one on the emotional subscale and the other on the functional subscale. The global question is scored and interpreted separately. The scores of all the items in each domain are summed and a mean score is calculated. The final score for each subscale is calculated by multiplying the calculated mean score by 20 with a final range from 0 to 100. The final score of the global question is also calculated in the same way. The higher the final score represents better functioning and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Raimond Wong, MD, Principal Investigator — McMaster University
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada